CLINICAL TRIAL: NCT02899585
Title: Expression of a Need of Implication for the Vulnerable Patient and His Adaptation
Acronym: EIVA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/27; 2014-A01386-41 (Other: ANSM)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Incurable Disease
Keywords: Palliative care
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Elaboration of the questionnaires
  Interventions: Other: Questionnaires
- Group B (Experimental): Patients taken care for more less than 6 days by the health care team palliatives EIVA and they eventual family caregiver. Score
  Interventions: Other: Questionnaires; Other: Score

INTERVENTIONS:
Other: Questionnaires
Other: Score
  Arms: Group B

SUMMARY:
The aim of the research is to detect prematurely vulnerable patients needing a global coverage in integrated care with a created and metrological validated score.

DETAILED DESCRIPTION:
The respect for the rights of the patients in palliative phase - having an evolutionary or terminal grave pathology - is a legal requirement since 1999, strengthened by the laws of April 4th, 2002 and April 22nd, 2005. Nevertheless, a lack of palliative approach persists, that is premature awareness of the necessity of a global approach, not exclusively centred on the specific therapeutics. The palliative approach remains rare and especially most of the time reduced in the last days of the life. The lack of distribution of the legal texts and insufficient training are among the main reasons. The lack of educational tools is probably also a major brake in a premature reflection.

Primary objective : to detect prematurely vulnerable patients needing a global coverage in integrated care with a created and metrological validated score.

Primary endpoint: capacity of the score to be discriminated (area under the curve) to find the patients who need or not a palliative approach

Secondary objectives:

* The measure of the relevance of the tests of quality of life, personality traits, level of information and anxiety depression to detect prematurely the vulnerable patients and/or their family caregivers who need an approach of palliative care in integrated care;
* The detail (date, nature of the event) of the various stages of their life course, during which the vulnerable patients needing a premature global care were taken care within the framework of such an approach, compared with their theoretical detection by the score of premature detection scale;
* The evaluation of the concordance between the patient score and the family caregiver score, if he participates in the research.

Secondary endpoints:

* The tests estimating the anxiety and the depression ( HAD (Hospital Anxiety and Depression) score), the personality and adaptation traits, Brief Cope;
* The quality of life tests EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire) and level of information EORTC INF-30 (Information-30) for the cancer patients;
* The deadline between detection by the score and effective global care
* The deadline between detection by the score and the cessation of the specific treatments
* The deadline between detection by the score and the death
* The patient and close scores obtained in the validation phase.

Methods: Prospective, controlled, nonrandomized study

Number of patients to include: 610 (maximum)

Duration: 36 months (32 inclusion months).

Number of participating centers: 1 center

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized with:

  * an evolutionary incurable disease;
  * Taken care for more than a month by the health care team palliatives EIVA (except for the last 200 patients, for whom the deadline extension of palliative care is lower that 6 days);
  * Benefiting of asocial scheme or claimant
  * Having signed the informed consent as well as his(her) family caregiver, if this one participates in the research.

The absence of family caregiver is not an exclusion criterion.

Exclusion Criteria:

* Patient:

  * Having difficulty of understanding of the French language
  * Having a life expectancy estimated unless one month
  * un controlled physical or psychic distress (anxiety and/or depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Capacity of the score to be discriminated (area under the curve) to find the patients who need or not a palliative approach | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Ferrand, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Arraras JI, Greimel E, Sezer O, Chie WC, Bergenmar M, Costantini A, Young T, Vlasic KK, Velikova G. An international validation study of the EORTC QLQ-INFO25 questionnaire: an instrument to assess the information given to cancer patients. Eur J Cancer. 2010 Oct;46(15):2726-38. doi: 10.1016/j.ejca.2010.06.118. Epub 2010 Jul 30. PMID 20674333
- [Result] Ferrand E, Robert R, Ingrand P, Lemaire F; French LATAREA Group. Withholding and withdrawal of life support in intensive-care units in France: a prospective survey. French LATAREA Group. Lancet. 2001 Jan 6;357(9249):9-14. doi: 10.1016/s0140-6736(00)03564-9. PMID 11197395
- [Result] Ferrand E, Jabre P, Vincent-Genod C, Aubry R, Badet M, Badia P, Cariou A, Ellien F, Gounant V, Gil R, Jaber S, Jay S, Paillaud E, Poulain P, Regnier B, Reignier J, Socie G, Tardy B, Lemaire F, Brun-Buisson C, Marty J; French Mort-a-l'Hopital Group. Circumstances of death in hospitalized patients and nurses' perceptions: French multicenter Mort-a-l'Hopital survey. Arch Intern Med. 2008 Apr 28;168(8):867-75. doi: 10.1001/archinte.168.8.867. PMID 18443263
- [Result] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Result] Greer JA, Pirl WF, Jackson VA, Muzikansky A, Lennes IT, Heist RS, Gallagher ER, Temel JS. Effect of early palliative care on chemotherapy use and end-of-life care in patients with metastatic non-small-cell lung cancer. J Clin Oncol. 2012 Feb 1;30(4):394-400. doi: 10.1200/JCO.2011.35.7996. Epub 2011 Dec 27. PMID 22203758
- [Result] Yoong J, Park ER, Greer JA, Jackson VA, Gallagher ER, Pirl WF, Back AL, Temel JS. Early palliative care in advanced lung cancer: a qualitative study. JAMA Intern Med. 2013 Feb 25;173(4):283-90. doi: 10.1001/jamainternmed.2013.1874. PMID 23358690
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Muller L, Spitz E. [Multidimensional assessment of coping: validation of the Brief COPE among French population]. Encephale. 2003 Nov-Dec;29(6):507-18. French. PMID 15029085